CLINICAL TRIAL: NCT06493903
Title: Physical and Mental Health Intervention for Black Adults With Knee Osteoarthritis: A Feasibility Study
Brief Title: Positive Minds Strong Joints for Knee Osteoarthritis
Acronym: PMSJ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Rheumatology Research Foundation (Other)
Responsible Party: Principal Investigator, Deepak Kumar, Associate Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7517
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Osteoarthritis, Knee
Keywords: chronic pain; depression; anxiety; exercise; cognitive behavioral therapy; Black adults
MeSH Terms: conditions — Osteoarthritis, Knee; Chronic Pain; Depression; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Positive Minds Strong Joints (Experimental): Participants will receive an individual mental health intervention through a zoom video-call once a week for 10 weeks and a community-based group exercise intervention once a week for 10 weeks.
  Interventions: Behavioral: Positive Minds, Strong Joints

INTERVENTIONS:
Behavioral: Positive Minds, Strong Joints — In this10-week physical and mental health intervention, participants will receive recommended exercise intervention and evidence-based mental health intervention for pain, depression and anxiety.

SUMMARY:
The aim of this research study is to test the feasibility of a physical and mental health intervention (Positive Minds, Strong Joints or PMSJ) for Black adults with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
In this feasibility study, at least 20 and up to 40 Black Adults will be enrolled to receive PMSJ intervention. Participants who will take part in this research study will be in it for about 26 weeks. Participants will receive a one-hour individual session of psychoeducation, mindfulness, and cognitive behavior therapy skills for 10 weeks via a HIPAA-protected zoom video-call or over the telephone. In addition, they will receive a community-based group exercise and pain education program once a week for 10 weeks. Participants will also continue to receive their usual care. Participants will be asked to take surveys at five time points (i.e.) before the start of the 10-week intervention (baseline visit), mid-way through the intervention (week 5), end of the 10-week intervention (post-intervention), 6 weeks after the intervention (week 16) and 12 weeks after the intervention (week 22). Brief surveys will also be completed weekly throughout the study. The surveys will be about pain, function, quality of life, mood, social support, sleep, etc. At baseline and post-intervention visits, all participants will also be asked to wear a small movement sensor on their lower back for 7 days of continuous movement and physical activity monitoring. During both of these 7-day periods, participants will complete a single remote assessment of their walking. Feasibility of the intervention will be determined post-intervention by outcome measures such as recruitment rate, retention rate, and adherence.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age≥50
* BMI ≤ 40 kg/m2
* Self-identify as Black (including African American)
* Knee pain ≥4/10 on a 11 numeric scale over the past week
* Scored 5 or more on either the Patient Health Questionnaire (PHQ-9) and/or the Generalized Anxiety Disorder 7-item Scale (GAD-7)
* Can speak and understand English at a sufficient level to understand the study procedures and informed consent
* Available for study duration
* Able to attend remote sessions

EXCLUSION CRITERIA

* Knee, hip or ankle replacement
* Intra-articular corticosteroid or hyaluronic acid knee injection within 3 months
* Knee surgery within past 6 months
* Currently receiving or received within 3-months any PT for knee OA
* Currently receiving or received within 3 months any mental health intervention (excluding pharmacologic treatments)
* Planning to initiate physical therapy for joint or low back pain in the next 3months
* Planning to initiate any mental health treatment (excluding pharmacologic treatments) in the next 1 month.
* Systemic inflammatory arthritis (e.g., rheumatoid arthritis)
* Neurologic conditions (e.g., stroke, Parkinson's disease, etc.)
* Contraindications to starting an exercise program.
* Suspected substance abuse
* Lack capacity to consent
* Pregnancy (self-report)
* Participation in another clinical trial for any joint or muscle pain
* Planning for a major surgery in the next 6 months
* Having high risk mental health symptoms (active suicidality, bipolar disorder, mania, psychosis, schizophrenia)
* Receiving chemotherapy or radiation therapy for cancer (except non-melanoma skin cancer)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Throughout the recruitment process
  Number of participants enrolled out of those screened
Retention | From the start of the study to end of the 10 week intervention
  Proportion of participants who complete patient-reported outcome surveys at 10 week timepoint
Attendance | During 10 weeks intervention period
  Proportion of participants that attended at least 80% of intervention sessions
Satisfaction with treatment | week 10 and week 22
  Custom 2-item (0-10 scale) to determine satisfaction with individual components of the intervention (i.e., Positive Minds, Strong Joints). There are 2 items and each item is scored separately. Higher scores for each item mean greater satisfaction for that dimension.
Participant Feedback | week 10 and week 22
  Custom survey asking the participants to provide feedback on a 5-point scale from very poor to excellent on various aspects of the intervention including content, interventionists, group aspects, overall rating, etc.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score | Baseline, week 5, week 10, week 16 and week 22
  Patient-reported outcome for knee pain and disability; a score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Patient Health Questionnaire 9-item | Baseline, week 5, week 10, week 16 and week 22
  9-item questionnaire assessing depression symptoms. Each question is scored from 0 to 3 where higher scores indicate higher frequency of experiencing depressive symptoms. Total score is the sum of individual item scores. Score range is 0-27. Higher total scores indicate greater severity of depression
Generalized anxiety 7-item scale | Baseline, week 5, week 10, week 16 and week 22
  It assesses anxiety symptoms. Each question is scored from 0 to 3 and the sum value of individual questions is the total score with range form 0-21. Higher total scores indicate greater severity of anxiety
Arthritis Self Efficacy Scale | Baseline, week 10, and week 22
  It measures confidence in one's capacity to function despite pain. Scores range from 1 (very uncertain) to 10 (very certain). It has three subscales of pain, function, and other symptoms calculated as average of items contributing to that subscale. Higher scores indicate greater self-efficacy to manage osteoarthritis.
Fear Avoidance Beliefs Questionnaire - Physical Activity | Baseline and week 10
  4-item questionnaire to determine how one's fear avoidance beliefs contributes to the cognitive/affective part of their knee pain. Each item is scored from 0 to 6. Total scores are summation of each item scores. Range is 0-24. Higher total scores indicate greater fear of physical activity
Pain Catastrophizing Scale | Baseline and week 10
  Questionnaire for a person's thought and feeling about pain. The questionnaire has 3 subscales namely rumination, magnification and helplessness. Each question is rated on a 5-point scale, from 0 (not at all) to 4 (always). It is scored by summing the ratings of its 13 items with a range of 0-52. Higher scores indicate greater pain catastrophizing tendencies in response to pain.
Trust in Medical Research Questionnaire | Baseline and week 10
  It assesses participants' trust in medical research. It includes items related to confidence in researchers, and the scientific process, rated on a 5 Likert scale (strongly disagree, disagree, neutral, agree and strongly agree) with a total score range of 0-48. Higher scores indicate greater trust in medical research
Multidimensional Scale of Perceived Social Support | Baseline and week 10
  It measures perceived social support from family, friends, and significant others. It consists of 12 items rated on a 7- Likert scale for a total score range from 12-84. Higher scores indicate greater perceived social support across various domains.
International Physical Activity Questionnaire | Baseline, week 10, week 22
  It assesses physical activity levels across diverse populations. The responses are converted into MET (Metabolic Equivalent of Task) minutes per week. The results can be continuous or categorized. For the categorized results, individuals' physical activity categorized as low, moderate and high
Patient-Reported Outcomes Measurement Information System-sleep | Baseline, week 10
  It is used to measure measures perceived sleep quality, difficulty in sleep and having enough and refreshing sleep. The 8 questions are rated on a 5-point scale. The scores are summed together with a raw score of from 8 to 40. The raw scores are then converted to standardized T-scores using conversion tables.
Patient Global Rating of Change | Week 10, Week 22
  This is a single item questionnaire with 15 options ranging from a very great deal worse to a very great deal better.
Numerical Rating Scale-nominated activity | Weekly from start of intervention to week 22
  average rating of knee pain from 0-10, where 0 represents no pain and 10 represents worst pain imaginable, in the past week in a nominated activity selected at baseline
Patient Global Assessment of Osteoarthritis | Weekly start of intervention to week 22
  It assesses participant's assessment of impact of osteoarthritis on their general health on a 0-100 scale. 0 is very poor and 100 is very well.
Adherence to exercise | Weekly from start of intervention to week 22
  This questionnaire is used to assess participants adhere to exercise. Participants document their engagement in unsupervised exercise throughout the week by noting minutes of exercise per day of the week
gait speed | Baseline and week 10
  A known distance of20-28 meters divided by time taken to walk this distance in m/s
Physical Activity Stages of change (short form) | Baseline and week 10
  It assesses participants readiness to engage physical activity. It consists of five stages which include Precontemplation, contemplation, preparation, action and maintenance.

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Requests will be considered on an individual basis

REFERENCES:
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Dillon CF, Rasch EK, Gu Q, Hirsch R. Prevalence of knee osteoarthritis in the United States: arthritis data from the Third National Health and Nutrition Examination Survey 1991-94. J Rheumatol. 2006 Nov;33(11):2271-9. Epub 2006 Oct 1. PMID 17013996
- [Background] Iversen MD, Schwartz TA, von Heideken J, Callahan LF, Golightly YM, Goode A, Hill C, Huffman K, Pathak A, Cooke J, Allen KD. Sociodemographic and Clinical Correlates of Physical Therapy Utilization in Adults With Symptomatic Knee Osteoarthritis. Phys Ther. 2018 Aug 1;98(8):670-678. doi: 10.1093/ptj/pzy052. PMID 29718472
- [Background] Jimenez DE, Cook B, Bartels SJ, Alegria M. Disparities in mental health service use of racial and ethnic minority elderly adults. J Am Geriatr Soc. 2013 Jan;61(1):18-25. doi: 10.1111/jgs.12063. Epub 2012 Dec 18. PMID 23252464
- [Background] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] McClendon J, Essien UR, Youk A, Ibrahim SA, Vina E, Kwoh CK, Hausmann LRM. Cumulative Disadvantage and Disparities in Depression and Pain Among Veterans With Osteoarthritis: The Role of Perceived Discrimination. Arthritis Care Res (Hoboken). 2021 Jan;73(1):11-17. doi: 10.1002/acr.24481. PMID 33026710
- [Background] Vaughn IA, Terry EL, Bartley EJ, Schaefer N, Fillingim RB. Racial-Ethnic Differences in Osteoarthritis Pain and Disability: A Meta-Analysis. J Pain. 2019 Jun;20(6):629-644. doi: 10.1016/j.jpain.2018.11.012. Epub 2018 Dec 10. PMID 30543951